CLINICAL TRIAL: NCT03748056
Title: Individually-targeted Incentives, Diet Quality, and Health Outcomes Among Adults
Brief Title: Targeted Food Incentives to Improve Diet Quality and Health Among Adults
Acronym: Smartcart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1240194-3; AWD05956 , Project 0006418 (Other Grant/Funding Number: Foundation for Food and Agricultural Research)
Record Dates: First submitted 2018-07-18; First posted 2018-11-20 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Diet Modification; Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted incentives arm (Experimental): The interventions received by the experimental group include: 1) weekly emails with targeted coupons for healthier products, 2) weekly emails with targeted nutrition education, and 3) and a nominal discount on grocery purchases for using their loyalty card
  Interventions: Behavioral: Targeted incentives; Behavioral: Nominal loyalty card discount and nutrition education
- Usual care arm (Active Comparator): The interventions included under "usual care" include 1) untargeted nutrition education, 2) occasional untargeted coupons for healthier products, and 3) a nominal discount on their grocery purchases for using their loyalty card. These interventions are only received by participants randomized to the usual care arm (rather than the entire population of shoppers), and will allow for testing whether targeting discounts and nutrition education improves the diet quality of purchases in comparison to untargeted approaches.
  Interventions: Behavioral: Nominal loyalty card discount and nutrition education

INTERVENTIONS:
Behavioral: Targeted incentives — Participants receiving individually-targeted incentives will receive weekly coupons for healthier foods that are informed by their purchase history, responses to behavioral and health questions, food preferences, and need for improvement in different categories
  Arms: Targeted incentives arm
Behavioral: Nominal loyalty card discount and nutrition education — All participants will receive a nominal discount on all groceries for using their loyalty card and nutrition education through weekly emails.

SUMMARY:
The purpose of this study is to test whether individual-level targeted price incentives for healthier foods can improve the diet quality of grocery purchases made by adults in comparison to a "one size fits all" approach. To test this, the investigators plan to implement a 8-month randomized controlled cross-over trial. The intervention group will receive a small discount for using their loyalty card and weekly coupons for healthier foods (e.g. fruits, vegetables, whole grains, lean meats and seafood, low-fat dairy) that are selected based on the individual's past purchase history, dietary preferences, their baseline diet quality, and their estimated likelihood of using the coupon. Individualized coupons will be automatically sent to customers' loyalty cards each week, and separate emails with appropriate nutrition education and information about the coupons will be sent to participants weekly. The control group will receive a small discount for using their loyalty cards during the first phase of the study (3-months), occasional untargeted coupons, and weekly emails with untargeted nutrition education. Following phase1, there will be a 2-month washout period, and then the intervention and control groups will cross over for the remaining 3-months of the study. The investigators will collect purchase data from all participants as well as food frequency questionnaires and other self-reported behavioral and health questions at baseline, after phase 1 completion, and after phase 2 completion. The investigators hypothesize that participants in the intervention group will meaningfully improve the overall quality of their food purchases (measured using the Grocery Purchase Quality Index-2016) as well as their overall diet quality (measured using the Healthy Eating Index 2010.

DETAILED DESCRIPTION:
A detailed description of Eligibility and outcome measures is entered elsewhere

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Speaks English
* Non-store employee
* Primary shopper in the household
* Purchases at least half of weekly groceries at supermarket
* Not pregnant or planning on becoming pregnant before April 2019

Exclusion Criteria:

* Younger than 18 years of age
* Does not speak English
* Employee at supermarket
* Pregnant or planning to become pregnant before April 2019
* Not primary shopper for household
* Purchases less than half of weekly groceries at supermarket

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Likelihood of purchasing targeted products | 3- 6- and 9-month changes within and between the intervention and control groups
  Within produce, whole grain cereals & breads, lean meats, low-fat dairy, and beverages, will look at the proportion of expenditures (i.e. percent of dollars) in those categories before and after the intervention between treatment and control group.
Grocery Purchase Quality Index (GPQI) 2016 | 3, 6- and 9-month changes in the GPQI-16 and its components within and between the intervention and control groups
  The GPQI is a validated measure for scoring the quality of household grocery purchases by comparing the percent spent within different food categories with recommended spending.
  https://utah.pure.elsevier.com/en/publications/the-grocery-purchase-quality-index-2016-an-innovative-approach-to

SECONDARY OUTCOMES:
Healthy Eating Index (HEI) -2010 for the primary shopper | 3, 6- and 9-month changes in the HEI-10 and its components within and between the intervention and control groups
  The HEI-10 is a validated measure of individual-level diet quality that measures compliance with US Dietary recommendations.
  https://www.ncbi.nlm.nih.gov/pubmed/24453128
Percent expenditures within targeted categories | 3, 6- and 9-month changes in percent spending in targeted categories within and between the intervention and control groups
  The investigators will compute the percent of shopping dollars people spend in fruits, vegetables, whole grains, dairy, lean meat, and seafood.
Self-reported height and weight used to compute body mass index (BMI) | 3, 6- and 9-month changes in BMI
  The investigators will compute body mass index from self-reported weight in pounds and height in inches (weight (lbs) * 703/height (in)/height (in)

OTHER OUTCOMES:
Self-reported food neophobia as an effect modifier on the primary and secondary outcomes | Baseline and 9-months
  The investigators will examine whether food neophobia modifies the effect of the intervention on the primary and secondary outcomes. Food neophobia was measured via 8 self-reported questions with a 5-point Likert scale ranging from completely disagree to completely agree. Responses will be summed, and higher scores reflect greater variety-seeking in eating experiences (i.e. less neophobia). We will test for an interaction between this continuous measure and the intervention on specified primary and secondary outcomes
Self-reported food literacy as an effect modifier on the primary and secondary outcomes | Baseline
  The investigators will examine whether food literacy modifies the effect of the intervention on the primary and secondary outcomes. Food literacy was measured using a 12-item questionnaire, with 4- and 5-point Likert type scales, with higher scores indicating greater food literacy.
Coupon proneness as an effect modifier on the primary and secondary outcomes | Baseline and 9-months
  The investigators will examine whether coupon proneness modifies the effect of the intervention on the primary and secondary outcomes. Coupon proneness was measured via a 22-item self-reported questionnaire with 7-point Likert scales. Higher scores indicate greater likelihood of using coupons.
Nutritional self-efficacy as a modifier on the primary and secondary outcomes | Baseline
  The investigators will examine whether nutritional self-efficacy modifies the effect of the intervention on the primary and secondary outcomes. Nutrition self-efficacy was measured via self-report using a 5-item scale with Likert responses (range 0-3) with higher scores indicating greater self-efficacy in nutritional domains.
Food security as a modifier on the primary and secondary outcomes | Baseline and 9-months
  The investigators will examine whether food security modifies the effect of the intervention on the primary and secondary outcomes. Household food security was assessed via a 6-item short form, with higher scores indicating greater food insecurity.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Vadiveloo, Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damsbo-Svendsen M, Frost MB, Olsen A. A review of instruments developed to measure food neophobia. Appetite. 2017 Jun 1;113:358-367. doi: 10.1016/j.appet.2017.02.032. Epub 2017 Mar 6. PMID 28268200
- [Background] VAN TRIJP HCM, STEENKAMP J-BEM. Consumers' variety seeking tendency with respect to foods: Measurement and managerial implications. Eur Rev Agric Econ. 1992;19(2):181-195. doi:10.1093/erae/19.2.181.
- [Background] Grea Krause C, Beer-Borst S, Sommerhalder K, Hayoz S, Abel T. A short food literacy questionnaire (SFLQ) for adults: Findings from a Swiss validation study. Appetite. 2018 Jan 1;120:275-280. doi: 10.1016/j.appet.2017.08.039. Epub 2017 Sep 11. PMID 28912107
- [Background] Lichtenstein, Ridgway, and Netemeyer. (1993) Price perception Scales. Handbook of Marketing Scales.
- [Background] University of Minnesota. Project EAT - Epidemiology & Community Health Research. http://www.sphresearch.umn.edu/epi/project-eat/#EAT3. Accessed June 14, 2018.
- [Background] Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. Am J Public Health. 1999 Aug;89(8):1231-4. doi: 10.2105/ajph.89.8.1231. PMID 10432912
- [Derived] Vadiveloo MK, Parker HW, Thorndike AN. Participant Characteristics Associated with High Responsiveness to Personalized Healthy Food Incentives: a Secondary Analysis of the Randomized Controlled Crossover Smart Cart Study. J Nutr. 2023 Jan 14;152(12):2913-2921. doi: 10.1093/jn/nxac197. PMID 36040345
- [Derived] Vadiveloo M, Guan X, Parker HW, Perraud E, Buchanan A, Atlas S, Thorndike AN. Effect of Personalized Incentives on Dietary Quality of Groceries Purchased: A Randomized Crossover Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2030921. doi: 10.1001/jamanetworkopen.2020.30921. PMID 33566105